CLINICAL TRIAL: NCT02601170
Title: Platelet-Rich Plasma Intra-Articular Injection in Treating Hemophilic Arthropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tsung-Ying Li, Attending physician, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-102-05-019
Record Dates: First submitted 2015-11-07; First posted 2015-11-10 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Hemophilia; Hemophilic Arthropathy
Keywords: Platelet Rich Plasma; Hemophilia; Hemophilic arthropathy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP Group (Experimental): single intra-articular injection of 2mL PRP (RegentKit-THT-1, RegenLab SA, Mont-sur-Lausanne, Switzerland)
  Interventions: Biological: Platelet-Rich Plasma Intra-Articular Injection
- HA Group (Active Comparator): five weekly intra-articular injections of 2.5 mL of hyaluronate sodium (ARTZDispo, Seikagaku Corporation Japan).
  Interventions: Drug: Hyaluronic Acid Viscosupplementation

INTERVENTIONS:
Biological: Platelet-Rich Plasma Intra-Articular Injection
  Arms: PRP Group
Drug: Hyaluronic Acid Viscosupplementation
  Arms: HA Group

SUMMARY:
Severe hemophilia is characterized by frequent and lifelong bleeding, with more than 60% of bleeds occurring into joints . Repeated joint bleeding leads to chronic synovitis, cartilage damage and bony destruction. Currently available treatment of hemophilic arthropathy, such as analgesics, NSAIDs, and hyaluronic acid (HA), are predominantly directed toward the symptomatic relief of pain and inflammation, but they do little to reduce joint cartilage degeneration.

Platelet-Rich Plasma (PRP) is a simple and minimally invasive method that provides a natural concentrate of autologous growth factors from the blood. This method is now being increasingly applied in clinical practice to treat musculoskeletal disorders, such as tendon repairment and osteoarthritis. To the best of our knowledge, no study applies PRP for arthropathy of knee joint in hemophilia patients. The aim of the study is to investigate the efficacy, safety and duration of benefit of single PRP injection versus five weekly intra-articular injections of HA in patients with hemophilic arthropathy of knee.

DETAILED DESCRIPTION:
Severe haemophilia is characterized by frequent and lifelong bleeding, with more than 60% of bleeds occurring into joints. Repeated joint bleeding leads to chronic synovitis, cartilage damage and bony destruction, which are associated with limitation of range of motion (ROM), pain, muscle atrophy, functional impairment, and poor quality of life. The knee, elbow, and ankle are the most commonly involved joints and arthropathy could worsen in adolescence or young adulthood. Hemophilic arthropathy is a multifactorial event and there is evidence to suggest that iron may play a major role with release of cytokines such as Interleukin ( IL)-1, IL-6, and tumour necrosis factor alpha (TNF-α) leading to chronic proliferative synovitis, hypervascularity, and progressive arthropathy. These effects on cartilage and subchondral bone are inflammatory and degenerative in nature and management of chronic hemophilic arthropathy is difficult.

Currently available drugs for the treatment of hemophilic arthropathy, such as analgesics, corticosteroids, nonsteroid and steroid anti-inflammatory drugs, and hyaluronic acid (HA), are predominantly directed toward the symptomatic relief of pain and inflammation, but they do little to reduce joint cartilage degeneration.

Platelet Rich Plasma (PRP) is a simple and minimally invasive method that provides a natural concentrate of autologous growth factors from the blood. This method is now being increasingly applied in clinical practice to treat musculoskeletal disorders, such as tendon repairment and osteoarthritis. Growth factors including platelet derived growth factor (PDGF), insulin growth factor (IGF), vascular endothelial growth factor, and transforming growth factor beta-1 are believed to be key components of PRP for structural repair. Although comparing PRP with other intra-articular and soft tissue injections has led to conflicting results, it seems that PRP has useful effects on healing and functional improvement of injured tissues. To the best of our knowledge, only one study applies PRP for arthropathy in haemophilia. Teyssler et al reported PRP could reduce pain of chronic ankle synovitis in hemophilia although the small sample size (n=6), short term follow-up and absence of a control group.

Hyaluronic acid (HA) has some role in joint mechanical support and its metabolic effects, which causes endogenous HA synthesis, stimulation of chondrocyte metabolism, synthesis of cartilage matrix components, and inhibition of chondrodegenerative enzymes, as well as inflammatory process. In 1994 Fernandez-Palazzi et al firstly used intra-articular HA injection for haemophiliacs with arthropathy and reported its beneficial effects in 2002. Recently, Carulli et al reported 27 haemophilic patients with a mean seven-year follow-up who had excellent results in terms of pain relief and functional improvement in the knee following treatment with HA injection. Viscosupplementation is a safe and effective therapeutic strategy in haemophilic arthropathy of knee in order to delay of surgery.

The aim of the study was to investigate the efficacy, safety and duration of benefit of single PRP injection versus five weekly intra-articular injections of HA in patients with haemophilic arthropathy of knee.

ELIGIBILITY:
Inclusion Criteria:

* hemophilia patients with hemophilic arthropathy of knee joints for at least 6 months
* painful (VAS ≥ 3) hemophilic arthropathy of knee joints after medication

Exclusion Criteria:

* presence of joint infections, any surgery on the joint in preceding 12 months
* intra-articular corticosteroid or HA injection within the past 6 months
* treatment with systemic steroids
* history of rheumatoid arthritis, or gouty arthropathy
* history of chicken or egg allergy
* presence of neoplasm
* use of non steroidal anti-inflammatory drugs in the 5 days before study
* platelet values < 100,000/mm3
* acute hemarthrosis
* paresis, or recent trauma.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- PRP Group: single intra-articular injection of 2mL PRP (RegentKit-THT-1, RegenLab SA, Mont-sur-Lausanne, Switzerland)
  Platelet-Rich Plasma Intra-Articular Injection
- HA Group: five weekly intra-articular injections of 2.5 mL of hyaluronate sodium (ARTZDispo, Seikagaku Corporation Japan).
  Hyaluronic Acid Viscosupplementation
Period: Overall Study
Arm/Group | PRP Group | HA Group
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRP Group | HA Group | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (2.3) | 38.8 (2.4) | 40.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Pain (Visual Analogue Scale) and Change From Baseline at 1, 2, 3 &6 Months
Description: The pain intensity will be evaluated subjectively on a visual analogue scale (0-10).
  Higher scores mean a worse outcome.
Time Frame: baseline, 1 month, 2 months, 3 months, 6 months
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | PRP Group | HA Group
Number analyzed (Participants) | 11 | 11
scores on a scale
  Baseline | 5.0 (0.6) | 4.1 (0.5)
  1 month | 2.5 (0.8) | 1.8 (0.5)
  2 months | 2.4 (0.8) | 1.6 (0.5)
  3 months | 2.5 (0.8) | 2.3 (0.6)
  6 months | 2.6 (0.7) | 3.4 (0.5)
Statistical Analysis 1: Comparison: PRP Group vs HA Group; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) From Baseline at 1, 2, 3 &6 Months
Description: It consists of 24 items: five pertaining to pain perception, two to stiffness, and 17 to physical function.
  Individual scores were then summed to form a raw score ranging from 0 (best) to 2400 (worst). Finally, WOMAC total score normalized between 0 (best) and 100 (worst).
Time Frame: baseline, 1 month, 2 months, 3 months, 6 months
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | PRP Group | HA Group
Number analyzed (Participants) | 11 | 11
scores on a scale
  Baseline | 38.3 (3.4) | 33.4 (5.5)
  1 month | 28.7 (3.7) | 19.1 (3.9)
  2 months | 27.3 (3.3) | 21.3 (3.7)
  3 months | 29.9 (3.9) | 27.1 (4.7)
  6 months | 29.4 (3.7) | 35.8 (5.0)

3. Secondary Outcome: Short Form-36 (SF-36) From Baseline at 1, 2, 3 &6 Months
Description: The SF-36 is a 36-item assessment tool that measures eight general health concepts including physical functioning, role limitation due to physical health problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems, and mental health. Individual scores were then summed to form a total score ranging from 0 (worst) to 100 (best). Higher scores mean a better outcome.
Time Frame: baseline, 1 month, 2 months, 3 months, 6 months
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | PRP Group | HA Group
Number analyzed (Participants) | 11 | 11
scores on a scale
  Baseline | 56.7 (5.3) | 54.7 (4.9)
  1 month | 62.8 (4.6) | 58.5 (5.0)
  2 months | 63.5 (4.1) | 63.5 (3.6)
  3 months | 61.7 (4.7) | 63.3 (3.1)
  6 months | 65.1 (3.7) | 58.3 (4.7)

4. Secondary Outcome: Ultrasonographic Synovial Thickness (mm) and Change From Baseline at 1, 2, 3 &6 Months
Description: Synovial thickness (mm) by ultrasonography were evaluated from the lateral, middle, and medial aspects of the anterior suprapatellar recess
Time Frame: baseline, 1 month, 2 months, 3 months, 6 months
Measure: Mean (Standard Error); unit: mm
Arm/Group | PRP Group | HA Group
Number analyzed (Participants) | 11 | 11
mm
  Baseline | 8.0 (1.3) | 6.9 (1.0)
  1 month | 7.1 (1.0) | 6.5 (1.2)
  2 months | 7.0 (1.3) | 6.1 (1.1)
  3 months | 7.2 (1.2) | 6.0 (1.1)
  6 months | 6.9 (1.0) | 6.0 (1.1)

5. Secondary Outcome: Synovial Hyperemia (Score) and Change From Baseline at 1, 2, 3 &6 Months
Description: Power Doppler assessment of the selected synovial sites was performed with settings standardized to a pulse repetition frequency of 700 Hz. The power Doppler gain was adjusted to a level just below the disappearance of artifacts under the bony cortex.14,15 The intensity of blood flow in the synovium was scored on a semiquantitative scale from 0-3 (grade 0, no intraarticular colour signal; grade 1, up to 3 color signals or 2 single and 1 confluent signal in the intraarticular area; grade 2, greater than grade 1 to <50% of the intraarticular area filled with color signals; grade 3, ≥50% of the intraarticular area filled with color signals)
Time Frame: baseline, 1 month, 2 months, 3 months, 6 months
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | PRP Group | HA Group
Number analyzed (Participants) | 11 | 11
scores on a scale
  Baseline | 1.0 (0.3) | 0.9 (0.2)
  1 month | 0.9 (0.3) | 0.4 (0.1)
  2 months | 0.3 (0.2) | 0.2 (0.1)
  3 months | 0.4 (0.2) | 0.3 (0.1)
  6 months | 0.3 (0.1) | 0.3 (0.1)

6. Secondary Outcome: Range of Motion (ROM, Degrees) From Baseline at 1, 2, 3 &6 Months
Time Frame: baseline, 1 month, 2 months, 3 months, 6 months
Measure: Mean (Standard Error); unit: degree
Arm/Group | PRP Group | HA Group
Number analyzed (Participants) | 11 | 11
degree
  Baseline | 92.3 (8.5) | 90.9 (8.3)
  1 month | 99.5 (7.6) | 91.8 (8.1)
  2 months | 102.3 (7.9) | 91.8 (8.1)
  3 months | 101.4 (7.8) | 91.8 (8.1)
  6 months | 100.9 (8.5) | 91.8 (8.1)

7. Secondary Outcome: Hemarthrosis From Baseline at 1, 2, 3 &6 Months
Description: Episode(s) of hemarthrosis in the previous one month
Time Frame: baseline, 1 month, 2 months, 3 months, 6 months
Measure: Mean (Standard Error); unit: episode (s)
Arm/Group | PRP Group | HA Group
Number analyzed (Participants) | 11 | 11
episode (s)
  Baseline | 0.5 (0.2) | 0.7 (0.2)
  1 month | 0.4 (0.2) | 0.4 (0.1)
  2 months | 0 (0) | 0.3 (0.1)
  3 months | 0.6 (0.3) | 0.3 (0.2)
  6 months | 0.4 (0.3) | 0.6 (0.2)

ADVERSE EVENTS:
Arm/Group | PRP Group | HA Group
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No